CLINICAL TRIAL: NCT02638090
Title: A Phase I/II Study of Pembrolizumab and Vorinostat in Patients With Immune Therapy Naïve and Immune Therapy Pretreated Stage IV NSCLC
Brief Title: Pembro and Vorinostat for Patients With Stage IV Non-small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18494
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Results first posted 2025-05-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: advanced lung cancer; immune therapy naive; immune therapy pre-treated; NSCLC; Stage IV lung cancer; pembrolizumab; vorinostat; immunogenicity
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Dose Escalation (Experimental): Level 1: Vorinostat 200mg by mouth (PO) Daily; Pembrolizumab 200 mg intravenously (IV) every (Q) 3 weeks.
  Level 2: Vorinostat 400 mg PO Daily; Pembrolizumab 200 mg IV Q3 weeks
  Interventions: Drug: Vorinostat; Drug: Pembrolizumab
- Phase Ib Expansion (Experimental): Pembrolizumab plus Vorinostat.
  Level 1: Maximum Tolerated Dose (MTD)
  Interventions: Drug: Vorinostat; Drug: Pembrolizumab
- Arm A: Pembrolizumab (Active Comparator): Pembrolizumab treatment only.
  Level 1: Pembrolizumab 200 mg Q3 wks
  Interventions: Drug: Pembrolizumab
- Arm B: Pembrolizumab plus Vorinostat (Active Comparator): Pembrolizumab plus Vorinostat treatment.
  Level 1: MTD
  Interventions: Drug: Vorinostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Vorinostat — Administered per treatment arm guidelines.
  Other Names: Zolinza
  Arms: Arm B: Pembrolizumab plus Vorinostat; Phase I Dose Escalation; Phase Ib Expansion
Drug: Pembrolizumab — Administered per treatment arm guidelines.
  Other Names: KEYTRUDA

SUMMARY:
The main purpose of this study is to see whether the combination of two drugs called pembrolizumab and vorinostat can help people with advanced lung cancer. Researchers also want to find out if the combination of pembrolizumab and vorinostat is safe and tolerable. This study will compare the effects of the combination of two drugs called pembrolizumab and vorinostat with the effects of pembrolizumab alone. The U.S. Food and Drug Administration (FDA) has approved pembrolizumab for use to treat a deadly skin cancer called melanoma and lung cancer and vorinostat to treat some forms of blood and lymph node cancers.

DETAILED DESCRIPTION:
A Phase I/Randomized Phase II clinical trial of pembrolizumab and vorinostat in Eastern Cooperative Oncology Group (ECOG) 0-1 patients with immune therapy naïve and immune therapy pretreated locally advanced or metastatic NSCLC who have progressed through one prior line of therapy.

The begins with a phase I dose escalation utilizing the modified continuous reassessment method (O'Quigley, Pepe, & Fisher, 1990). This would be followed by a phase I expansion at the maximum tolerated dose (MTD) in 18 NSCLC patients who have been previously treated with anti-PD-1 or anti-PD-L1 therapy. In parallel, a separate phase II arm will randomize 70 patients to a pembrolizumab alone group and a pembrolizumab plus vorinostat group.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Have archival tissue where available. Those participants enrolled on the phase 1 escalation trial where archival tissue is not available will undergo a fresh biopsy where clinically feasible after discussion with the sponsor.
* In addition, participants enrolled on the phase 1 dose escalation, phase 1 expansion or Phase II trial must be willing and able to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
* Randomized Phase II: Tumor proportional score of PD-L1 ≥1%.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function.
* Have a histologic or cytologic diagnosis of Stage IV non-small cell lung cancer (NSCLC).
* Phase I/IB (Pre-treated): Have progression from at least one prior line of therapy. Maintenance therapy following platinum doublet-based chemotherapy is not considered as a separate regimen of therapy. Participants who received platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, and developed recurrent (local or metastatic) disease within 6 months of completing therapy are eligible for these arms. Participants with recurrent disease ≥ 6 months after completing a platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, who also subsequently progressed during or after a systemic regimen given to treat the recurrence, must have received another treatment in the first-line metastatic setting.
* Randomized Phase II: Be treatment naïve in the stage IV setting, with the exception of participants whose tumors harbor an activation mutation (including but not limited to EGFR, ALK, ROS1) and were previously treated with targeted therapy. Participants who received platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, and developed recurrent (local or metastatic) disease < 6 months of completing therapy are ineligible for this arm. Subjects with recurrent disease ≥ 6 months after completing a platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, who also subsequently progressed during or after a systemic regimen given to treat the recurrence, are eligible for this arm.
* Females of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* Males should agree to use an adequate method of barrier contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating in and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at doses ≥ 10 mg prednisone or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Participants are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if >= 10 mg/day prednisone equivalents. A brief course (≤28 days) of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Has a known history of tuberculosis (TB) Disease (Mycobacterium tuberculosis).
* Hypersensitivity to pembrolizumab, vorinostat or any of its excipients.
* Participants enrolled on the phase II randomized trial, who have had prior treatment with a PD1 or PDL1 inhibitor, anti-CTLA 4 antibody or any other antibody or drug that specifically targets immune checkpoint pathway (i.e. not "immune therapy naïve"). -Note: For those enrolled in the phase I dose escalation, prior use of a PD1 or PDL1, anti-CTLA4 antibody or any other antibody or drug that specifically targets immune checkpoint pathway is allowed. For those enrolled in the phase IB, prior use of a PD1 or PDL1, anti-CTLA4 antibody or any other antibody or drug that specifically targets immune checkpoint pathway is required. For all participants in all phases, prior use of a vaccine for treatment of cancer is allowed.
* Participants enrolled in the phase Ib expansion who have never previously been treated with a PD1 or PDL1 inhibitor, anti-CTLA 4 antibody or any other antibody or drug that specifically targets immune checkpoint pathway in the past (i.e. not "pre-treated").
* Participants who have received thoracic radiation >30Gy within 6 months of the first dose of pembrolizumab.
* Patients taking any HDACi other than vorinostat.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy with 3 weeks, or targeted small molecule therapy or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Patients with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: Patients with any grade alopecia are an exception to this criterion and may qualify for the study.
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Previously treated brain metastases may be an exception if stable and specific other criteria are met.
* Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Has an active infection requiring systemic therapy.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has a history of, or any evidence of active non-infectious pneumonitis that required or requires steroids.
* Has evidence of interstitial lung disease
* Has a history of symptomatic (NYHA class II-IV) heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1- Dose Level 1: Level 1: Vorinostat 200mg by mouth (PO) Daily; Pembrolizumab 200 mg intravenously (IV) every (Q) 3 weeks.
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
- Phase I - Dose Level 2: Level 2: Vorinostat 400 mg PO Daily; Pembrolizumab 200 mg IV Q3 weeks
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
- Phase Ib Expansion: Pembrolizumab plus Vorinostat.
  Level 1: Maximum Tolerated Dose (MTD)
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
- Arm A: Pembrolizumab: Pembrolizumab treatment only.
  Level 1: Pembrolizumab 200 mg Q3 wks
  Pembrolizumab: Administered per treatment arm guidelines.
- Arm B: Pembrolizumab Plus Vorinostat: Pembrolizumab plus Vorinostat treatment.
  Level 1: MTD
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
Period: Overall Study
Arm/Group | Phase 1- Dose Level 1 | Phase I - Dose Level 2 | Phase Ib Expansion | Arm A: Pembrolizumab | Arm B: Pembrolizumab Plus Vorinostat
Started | 5 | 9 | 20 | 40 | 46
Completed | 4 | 9 | 20 | 40 | 43
Not Completed | 1 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Dose Level 1: Level 1: Vorinostat 200mg by mouth (PO) Daily; Pembrolizumab 200 mg intravenously (IV) every (Q) 3 weeks.
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase Ib Expansion | Arm A: Pembrolizumab | Arm B: Pembrolizumab Plus Vorinostat | Total
Number analyzed (Participants) | 5 | 9 | 20 | 40 | 46 | 120
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 82] | 66 [53 to 80] | 68 [38 to 80] | 69 [47 to 86] | 68 [44 to 87] | 68 [38 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 7 | 16 | 24 | 51
  Male | 3 | 7 | 13 | 24 | 22 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 5 | 8 | 20 | 37 | 43 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 4 | 7
  White | 4 | 8 | 19 | 38 | 41 | 110
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 20 | 40 | 46 | 120

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose (MTD) corresponding to a risk of dose limiting toxicity (DLT) occurring in 30% of patients. DLTs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.03). A DLT will be defined as any Grade 3 or higher toxicity that occurs during the DLT evaluation period. Toxicity that is clearly and directly related to the primary disease or to another etiology is excluded from this definition.
Time Frame: Up to 12 months
Measure: Number; unit: Milligrams of Vorinostat
Groups:
- Phase I Dose Escalation: Level 1: Vorinostat 200mg by mouth (PO) Daily; Pembrolizumab 200 mg intravenously (IV) every (Q) 3 weeks.
  Level 2: Vorinostat 400 mg PO Daily; Pembrolizumab 200 mg IV Q3 weeks
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
Arm/Group | Phase I Dose Escalation
Number analyzed (Participants) | 13
Milligrams of Vorinostat | 400

2. Secondary Outcome: Phase II: Progression Free Survival (PFS) Per Treatment Arm
Description: PFS will be measured from the start of treatment with pembrolizumab and vorinostat until the documentation of disease progression or death due to any cause, whichever occurs first. Progression: One or more of the following must occur: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Pembrolizumab | Arm B: Pembrolizumab Plus Vorinostat
Number analyzed (Participants) | 40 | 46
Months | 4.5 [2.1 to 9.3] | 4.3 [2.8 to 9.4]

3. Other Pre Specified Outcome: Phase II: Objective Response Rate (ORR) Per Treatment Arm
Description: Complete response (CR) or partial response (PR) based on modified Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1. The ORR will be estimated by calculating the proportion of participants who achieve OR; the 80% confidence interval (CI) and 95% CI for the OR rate will be estimated using the exact binomial distribution. CR: Complete disappearance of all target and non-target lesions (exception: lymph nodes mentioned below). No new lesions. No disease related symptoms. Any lymph nodes (target or non-target) must have reduction in short axis to < 1.0 cm. All disease must be assessed using the same technique as baseline. PR: Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: Up to 2 years
Measure: Number; unit: Percentage of Participants with OR
Arm/Group | Arm A: Pembrolizumab | Arm B: Pembrolizumab Plus Vorinostat
Number analyzed (Participants) | 40 | 43
Percentage of Participants with OR | 28 | 41

ADVERSE EVENTS:
Time Frame: All adverse events are recorded from C1D1 and for up to 2 years
Groups:
- Phase I Dose Escalation - Level 1: Level 1: Vorinostat 200mg by mouth (PO) Daily; Pembrolizumab 200 mg intravenously (IV) every (Q) 3 weeks.
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
- Phase I Dose Escalation - Level 2: Level 2: Vorinostat 400 mg PO Daily; Pembrolizumab 200 mg IV Q3 weeks
  Vorinostat: Administered per treatment arm guidelines.
  Pembrolizumab: Administered per treatment arm guidelines.
Arm/Group | Phase I Dose Escalation - Level 1 | Phase I Dose Escalation - Level 2 | Phase Ib Expansion | Arm A: Pembrolizumab | Arm B: Pembrolizumab Plus Vorinostat
All-Cause Mortality (participants affected / at risk) | 5/5 | 9/9 | 18/20 | 35/40 | 40/46
Serious Adverse Events (participants affected / at risk) | 4/5 | 3/9 | 14/20 | 16/40 | 26/46
Other Adverse Events (participants affected / at risk) | 5/5 | 8/9 | 20/20 | 40/40 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Escalation - Level 1 (N=5) | Phase I Dose Escalation - Level 2 (N=9) | Phase Ib Expansion (N=20) | Arm A: Pembrolizumab (N=40) | Arm B: Pembrolizumab Plus Vorinostat (N=46)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Alcohol intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Non-cardiac chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Escalation - Level 1 (N=5) | Phase I Dose Escalation - Level 2 (N=9) | Phase Ib Expansion (N=20) | Arm A: Pembrolizumab (N=40) | Arm B: Pembrolizumab Plus Vorinostat (N=46)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 7 (12) | 8 (10) | 27 (32)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 8 (10) | 5 (5) | 24 (32)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0) | 9 (9) | 2 (2) | 12 (14)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (2) | 6 (6) | 5 (5) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 7 (8)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (3) | 6 (8) | 9 (13) | 10 (11) | 21 (30)
Pain (General disorders) | 1 (2) | 3 (4) | 8 (10) | 13 (17) | 10 (17)
Fever (General disorders) | 0 (0) | 2 (3) | 5 (7) | 1 (1) | 6 (6)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 7 (10)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 4 (4)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 3 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Localized edema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 6 (10) | 13 (14) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 9 (9) | 8 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 9 (14) | 6 (6)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (6) | 5 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 10 (16)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 8 (10) | 7 (8) | 17 (22)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 8 (17)
Hyponatremia (Metabolism and nutrition disorders) | 1 (6) | 1 (1) | 5 (10) | 4 (6) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alcohol intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (17) | 5 (5) | 7 (13) | 4 (8) | 12 (20)
Weight loss (Investigations) | 2 (3) | 1 (1) | 5 (7) | 3 (4) | 4 (6)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 4 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 1 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (6) | 1 (3) | 3 (4)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (9) | 6 (8) | 8 (8)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 6 (7) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (6)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 6 (7)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 6 (7) | 1 (1) | 9 (10)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 6 (7)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 6 (7)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 2 (3)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 4 (4) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (8) | 7 (10) | 6 (8) | 9 (18)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 5 (5)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (6) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (5) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 3 (4)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT02638090/Prot_SAP_000.pdf